CLINICAL TRIAL: NCT05908656
Title: Implementation and Evaluation of a Rare Disease Algorithm to Identify Persons at Risk of Gaucher Disease Using Data From Electronic Health Records (EHRs) in the United States
Brief Title: Implementation and Evaluation of a Rare Disease Algorithm to Identify Persons at Risk of Gaucher Disease Using Data From Electronic Health Records (EHRs) in the United States (Project Searchlight)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PIR17206; U1111-1280-8450 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with electronic health records suggestive of Gaucher disease (Other)
  Interventions: Procedure: Investigational procedure

INTERVENTIONS:
Procedure: Investigational procedure — Subjects that consent will have a single blood draw either via a finger stick or via venous blood draw (blood will be placed on a 5 spot blood card) used to determine whether they have Gaucher Disease or ASMD

SUMMARY:
This is a three-phase study comprising both retrospective and prospective components, as follows:

Phase I: Deployment of Rare Disease Algorithm:

A diagnostic screening algorithm was developed using advanced analytical methods to identify patients who have an increased likelihood of having Gaucher disease. This tool will be applied to a health system's electronic health records (EHR).

The top 50 active patients per healthcare system will be identified as "highly ranked by the RDA" and moved to Phase II. As three to four healthcare systems are expected to participate in this study, between 150 to 200 persons are expected to be identified and included in Phase II.

Phase II: Retrospective review of medical records of highly ranked persons: The listing of persons highly-ranked by the RDA from phase I will be forwarded to the study team within each participating healthcare system. After reviewing the RDA reports and medical records of each highly ranked person, study site personnel will determine eligibility for Phase III based on the relevant selection criteria listed in the section below.

Phase III: Prospective diagnostic testing: Eligible persons (or their parent/guardian) from Phase II will be contacted and asked to provide consent for inclusion into the study. After consent is received, blood samples will be collected and sent for Gaucher diagnostic testing. Because of overlap in clinical symptoms between Gaucher disease and acid sphingomyelinase deficiency (ASMD), patients will also receive diagnostic testing for ASMD. Results will be shared with study site personnel, who will subsequently inform the study subject (and/or their parent/guardian, where appropriate) of results. It is anticipated that participation of a typical subject will be less than 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Phase I (Model Deployment): All persons within the EHRs of the selected IDNs will be included in this stage.
* Phase II (Case Ascertainment): The 150 to 200 persons with the highest RDA values (i.e., 50 per healthcare system) who are active (any documented interaction with the healthcare system in the previous 18 months) will be included in this stage.
* Phase III (Diagnostic Testing): The subset of persons from Phase II who: (1) have not been diagnosed with GD or ASMD, and (2) have not had GD and ASMD conclusively ruled out, will be asked to provide consent to undergo diagnostic testing. Individuals who meet these criteria and who provide written informed consent (or those whose parents/guardians provide consent as appropriate) will be included in this stage.

Exclusion Criteria:

* There are no exclusion criteria for Phase I or Phase II.
* Phase III (Diagnostic Testing):

  * Patient is unable/unwilling to provide informed consent for diagnostic testing, or
  * Patient is no longer under the care of the IDN

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
The proportion of persons with GD (including those with GD identified in Phase II and those previously undiagnosed who subsequently test positive for GD in Phase III) out of all persons highly ranked by the RDA | Up to 3 months
The proportion of previously undiagnosed persons highly ranked by RDA who subsequently test positive for GD out of persons with GD identified in Phase II and III | Up to 3 months

SECONDARY OUTCOMES:
Characteristics include demographic information, alternative and concomitant diagnoses, treatments, and patterns of provider visits for the previously listed subgroups | Up to 3 months
Relationship between RDA scores and the diagnostic yield; descriptive analyses including confusion matrices | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - University of Florida 655 W 8th St- Site Number : 8400003, Gainesville, Florida
  - Metropolitan Hospital Center- Site Number : 8400001, New York, New York
  - Aurora Research Institute LLC- Site Number : 8400002, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org